CLINICAL TRIAL: NCT07206420
Title: Balancing Acts: Impact of Medical Education on the Health and Lifestyle of Aspiring Physicians, a Cross-Sectional Study
Brief Title: Balancing Acts: Impact of Medical Education on the Health and Lifestyle of Aspiring Physicians
Status: Completed | Type: Observational
Sponsor: Nishtar Medical University (Other)
Responsible Party: Principal Investigator, Fatima Naveed, MBBS student, Nishtar Medical University
Other Study IDs: 8974/NMU
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-09

CONDITIONS: Diet Habits; Sleep Hygiene; Physical Activities
Keywords: Medical education; Medical students; Health; Stress; Diet; Physical activity; Cross-Sectional Study
MeSH Terms: conditions — Feeding Behavior; Sleep Hygiene; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Medical Students: Undergraduate medical students enrolled at Nishtar Medical University, Multan, who completed a structured questionnaire assessing lifestyle, health behaviors, and the impact of medical education.

SUMMARY:
This cross-sectional study explored the impact of medical education on the health and lifestyle behaviors of undergraduate medical students at Nishtar Medical University, Multan. Medical training is known to be academically and emotionally demanding, which can significantly influence students' physical activity, nutrition, sleep, and mental well-being.

Data were collected through a structured, self-administered questionnaire distributed to medical students across different years of study. The survey assessed lifestyle domains including diet, exercise, sleep patterns, stress, and coping mechanisms. Demographic details and academic year were also recorded.

The primary objective was to evaluate the association between the intensity of medical education and students' overall health and lifestyle. Findings aim to provide insight into how medical training environments shape future physicians' personal health practices and to identify potential areas for institutional support and wellness interventions.

ELIGIBILITY:
Inclusion Criteria:

* All Undergraduate medical students

Exclusion Criteria:

* Graduate medical students and doctors

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Undergraduate medical students enrolled at Nishtar Medical University, Multan, who completed a structured questionnaire assessing health behaviors, lifestyle, and the impact of medical education on well-being.
Sampling Method: Non-Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2025-05-12 (Actual); Primary Completion 2025-07-20 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Lifestyle and health behaviors of medical students | Baseline (single assessment at study enrollment) (cross-sectional).
  Lifestyle domains including diet, physical activity, sleep patterns, stress levels, and coping strategies were assessed using a structured self-administered questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Fatima Naveed, Multan, Pakistan

IPD SHARING:
Plan to Share IPD: No